CLINICAL TRIAL: NCT00837980
Title: Investigation of the Role of Functional Imaging in Characterising Radiotherapy Target Volumes and Assessing Disease Response in Patients Undergoing Chemoradiation for Head and Neck Cancer (HNC)
Brief Title: Functional Imaging in HNC Undergoing Chemoradiation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Dr Kate Newbold/ Chief Investigator, Royal Marsden Hospital NHS Foundation Trust
Other Study IDs: CCR3123
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer; DW MRI; PET; DCE MRI; functional imaging; IMRT
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to generate a library of functional imaging and anatomical imaging for patients with head and neck cancers for evaluation of new radiotherapy strategies and planning techniques including IMRT. Secondary aims would be to observe the changes in the cancers as the treatment progresses as well as to define the biologically most active part of the tumor (biological target volume) which could be given more intensive treatment. Tumor volumes seen on different imaging modalities will be compared with a hope of finding an optimal imaging methodology for accurate visualization of the head and neck cancers

DETAILED DESCRIPTION:
Adult patients who have a head and neck cancer and are planned to receive chemotherapy and radiotherapy will be invited to participate in the study. Patients who are not in very good health, have diabetes or kidney failure will not be considered for the study. Also patients who can not undergo MRI scan or are allergic to contrast injection given prior to the scan or have had any other form of cancer (except skin cancer) will also be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* patients with histologically proven head and neck cancer, planed for chemotherapy and radiotherapy
* age more than 18 years
* patient willing to participate and has signed a consent form
* patients in good physical status (WHO performance status 0-2)

Exclusion Criteria:

* patients in poor health (WHO performance status >2)
* patients with any other cancer apart from skin cancer
* patients with contraindications to MRI scan and IV contrast
* diabetic patients
* patients with renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who have a head and neck cancer and are planned to receive chemotherapy and radiotherapy will be invited to participate in the study. Patients who are not in very good health, have diabetes or kidney failure will not be considered for the study. Also patients who can not undergo MRI scan or are allergic to contrast injection given prior to the scan or have had any other form of cancer (except skin cancer) will also be excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-11 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
the number of patients completing the study protocol and adding to the library of images to be used for evaluation of new radiotherapy strategies and planning techniques including IMRT

SECONDARY OUTCOMES:
the ability to define a biological target volume in all the patients
to compare the volumes defined by the conventional imaging to the functional imaging
to measure changes in the volume of the disease with diff

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom